CLINICAL TRIAL: NCT06700876
Title: Evaluation of Interferon-gamma Release Assays, Symptom Screening and Chest Radiograph for Detection of Subclinical Tuberculosis of End-stage Kidney Disease and Kidney Transplant Recipients in Thailand
Brief Title: Evaluation of IGRA, Symptoms and Chest Radiograph for Subclinical TB Detection in ESRD and KT
Status: Recruiting | Type: Observational
Sponsor: Mahidol University (Other)
Collaborators: National Research Council of Thailand (Other Government)
Responsible Party: Principal Investigator, Punnee Pitisuttithum, Professor, Mahidol University
Other Study IDs: NRCT9-5
Record Dates: First submitted 2024-10-07; First posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Tuberculosis (TB); End-Stage Kidney Disease
Keywords: Subclinical Tuberculosis; Interferon gamma release assays; End-stage Kidney Disease; Detection of Subclinical Tuberculosis; Tuberculosis; IGRAs
MeSH Terms: conditions — Tuberculosis; Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood for IGRAs, Sputum MTB/RIF Xpert (Only the subject whose blood for IGRAs results are positive )
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 160 End-stage renal disease patients: End-stage renal disease on renal replacement therapy (hemodialysis or peritoneal dialysis) or status-post-living donor or deceased donor kidney transplantation aged more than or equal 18 years

SUMMARY:
This is an observational study among approximately 160 end-stage renal disease patients on renal replacement therapy and post-living donor or deceased donor kidney transplant recipients. Investigators aim to assess the proportion of positive IGRA associated with symptom development, sputum Xpert MTB/RIF assay, and chest radiograph to define latent TB infection and subclinical TB among ESKD and renal transplant patients.

DETAILED DESCRIPTION:
Patients with chronic kidney disease and end-stage kidney disease (ESKD) are at risk of developing tuberculosis and are often delayed in diagnosis. Herein, investigators aim to assess the proportion of positive IGRA associated with symptom development, sputum Xpert MTB/RIF assay, and chest radiograph to define latent TB infection and subclinical TB among ESKD and renal transplant patients.

ELIGIBILITY:
Inclusion Criteria:

1. End-stage renal disease on renal replacement therapy (hemodialysis or peritoneal dialysis) or status-post-living donor or deceased donor kidney transplantation
2. Aged more than or equal 18 years

Exclusion Criteria:

1. Positive PPD test or a previously documented positive PPD
2. Active pulmonary or extrapulmonary tuberculosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: End-stage renal disease on renal replacement therapy (hemodialysis or peritoneal dialysis) or status-post-living donor or deceased donor kidney transplantation aged more than or equal 18 years
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2024-08-06 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
1.The number of participants with positive IGRAs among end-stage kidney disease and kidney transplant patients | A prospective cohort study with following up period 2 years
  The number of participants with positive IGRAs among end-stage kidney disease patients and kidney transplant patients
2. The number of participants with latent TB and active TB among end-stage kidney disease and kidney transplant patients during the 2-year follow-up defined by: | A prospective cohort study with following up period 2 years
  1. Latent TB: a state of persistent immune response to stimulation by Mycobacterium tuberculosis antigens (positive IGRA) with no evidence of clinically manifest active TB
  2. Active TB: a disease in someone infected with Mycobacterium tuberculosis. It is characterized by signs or symptoms of active disease, or both, and is distinct from latent TB infection, which occurs without signs or symptoms of active disease

CONTACTS AND LOCATIONS:
Overall Officials: Punnee Pitisuttithum, Prof. E., Study Chair — Vaccine Trial Centre, Faculty of Tropical Medicine, Mahidol University
Locations (1):
- Vaccine Trial Centre, Faculty of Tropical Medicine, Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No